CLINICAL TRIAL: NCT05808959
Title: The Effect of Structured Education on Sexual Function and Sexual Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Hatice ÖNER CENGİZ, Assist. Prof., Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HONERCENGIZ
Record Dates: First submitted 2023-03-17; First posted 2023-04-12 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Arthropathy of Hip; Sexuality; Orthopedic Disorder
MeSH Terms: conditions — Sexuality; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education group (Experimental): Structured training on sexual health will be given to patients in this group. After the discharge training given at the clinic in the postoperative period, the participants will be given structured training on sexual health. It is anticipated that the training will take approximately 30 minutes. Immediately after the training, feedback will be received from the patient through a question-answer activity, and areas that are not understood will be repeated. It is thought that the training will take approximately 45-60 minutes in total.
  Interventions: Behavioral: Education group
- Control group (No Intervention): The clinic's routine discharge training will be applied to the participants in the control group.

INTERVENTIONS:
Behavioral: Education group — After the discharge training given at the clinic in the postoperative period, the participants will be given structured training on sexual health.
  Arms: Education group

SUMMARY:
An active sex life has an important place for the quality of life and is closely related to the increase in the general health level. In this context, a healthy sexual life after TKA surgery can contribute to the general quality of life of the patients. In the pre-TKA period, the sexual activity of female patients was found to be impaired more than men, the relationship between spouses was significantly affected negatively, and in the post-TKA period, general sexual recovery was significantly delayed in female patients compared to men. From this perspective, it is clear that pre- and post-TKA sexual counseling is important when preparing a balanced resumption of sexual activity in female patients after TKA. However, in clinical practice, patients may hesitate to talk about sexual life, and orthopedists and nurses often ignore this.

DETAILED DESCRIPTION:
Total Hip Arthroplasty (TKA) is a successful and major treatment modality that provides pain reduction/relief, functional recovery and increase in quality of life in patients with knee osteoarthritis and osteonecrosis (Turhan and Büyük 2022, Yamagami et al. 2021, Lei et al. 2019). The indication for TKA is increasing, especially in young patients with high functional expectations and who are sexually active (Kurtz et al. 2014). The World Health Organization (WHO) sexual health is "…a state of physical, emotional, mental and social well-being in relation to sexuality; it is not just the absence of disease, dysfunction, or disability." It has been defined as an important area of quality of life (WHO 2006). An active sex life has an important place for the quality of life and is closely related to the increase in the general health level. In this context, a healthy sexual life after TKA surgery can contribute to the general quality of life of patients (Neonakis et al 2020). Interruption or forcing of sexual life for a long time in the osteoarthritis process can also increase the expectations of patients from TKA intervention. However, after TKA, patients may limit themselves sexually, especially due to the fear of dislocation (Pritchett 2017, Yoon et al. 2013). It is clear that pre- and post-TKA sexual counseling is important when preparing for a balanced resumption of sexual activity in female patients after THA (Neonakis et al 2020). However, in clinical practice, patients may hesitate to talk about sexual life, and orthopedists and nurses often ignore this (Charbonnier et al. 2014, Peter et al. 2011). In one study, most of the patients could not get information about sexual activity after TKA and did not consult a doctor because of the specificity of the subject (Yoon et al. 2013), whereas in another study, only 17% of the patients received information about the onset of sexual activity and risky positions after surgery (Laffosse et al. 2008) were determined. However, some changes should be made in the sexual activities of patients after TKA intervention. Permissible sexual position after TKA differs according to gender, the approach used and the time after surgery. For this reason, it is very important for patients to receive an individualized education on sexual life for their postoperative sexual health (Neonakis et al. 2020). However, no study has been found in the literature evaluating the effectiveness of any training given to patients undergoing TKA in the pre- or postoperative period. In the light of this information, the aim of the study is to determine the effect of structured education on sexuality on sexual function and quality of sexual life in female patients undergoing TKA.

Method This single-center, randomized controlled trial Participants and Sample The population of the study will be female patients who underwent TKA in the clinic where the study will be conducted. G*Power (version 3.1.9.4) analysis was performed to determine sample size. it was planned to include 34 patients in total, 17 patients in each group.

Education Group; Their spouses will also participate in the structured sexual health education to be given to the women included in the training group and they will give their consent. Within the scope of the training, the definition of total hip replacement, the importance of sexual health, the definition of sexual intimacy, the ways of sexual intimacy, the general precautions that the patient should pay attention to in sexual life after TKA, the positions that should not be used during sexual intercourse in the early and late postoperative period, in the early postoperative period and In the late period, positions that can be used during sexual intercourse will be trained. It is thought that the training will take approximately 45-60 minutes in total.

Control Group; The participants in the control group will be given routine care of the clinic. Data Collection The data of the patient will be collected by the researchers face-to-face and through telephone interviews, using the Patient Sociodemographic and Medical Data Form, Female Sexual Function Questionnaire Index, Sexual Life Quality Scale-Female (CYQQ-F), Visual Analogue Scale (VAS).

Evaluation of Research Data SPSS 22.0 (IBM Corp., Armonk, NY) package program will be used in the evaluation of the data obtained from the research. Descriptive statistics will be presented as numbers, percentages, mean±standard deviation (SD), and median (min-max) values. Fisher's Exact Test or Pearson chi-square test will be used in the analysis of relationships between categorical variables. In the normality test, Shapiro Wilks test will be used when the number of samples in the group is less than 50, and Kolmogorov-Smirnov test will be used when it is large. In the analysis of the changes in the scores over time, the Kruskal Wallis test will be used if the measurements do not comply with the normal distribution, and the ANOVA test will be used if the measurements comply with the normal distribution. In the analysis of the difference between the scores of the two groups, the Mann-Whitney U test will be used if it does not fit the normal distribution, and the Student's t test will be used if it does. The reliability coefficient of the scales used in the study will be determined by calculating the Cronbach alpha coefficient. P values less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* >18-<65 years old,
* have no barriers to communicating,
* able to understand and speak Turkish,
* sexually active before and after TKA,
* with her husband,
* patients without sexual dysfunction will be included.

Exclusion Criteria:

* having a history of spinal surgery,
* having cancer,
* having a psychological or gynecological/urological disease, Exclusion criteria from the study;
* developing surgical site infection after TKA,
* do not complete the study,
* developing any complications during the working process,
* patients who lost their lives during the study will be excluded.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Sexual function-first evaluation | before surgery
  Sexual function will be evaluated 4 times in the perioperative period.Data will be collected with the Female Sexual Function Questionnaire Index. The highest score that can be obtained from the scale is 45, and as the total score decreases, it is considered as a decrease in sexual function.
Sexual function-second evaluation | 1 month after surgery
  Sexual function will be evaluated 4 times in the postoperative period.Data will be collected with the Female Sexual Function Questionnaire Index. The highest score that can be obtained from the scale is 45, and as the total score decreases, it is considered as a decrease in sexual function.
Sexual function-third evaluation | 3 month after surgery
  Sexual function will be evaluated 4 times in the postoperative period.Data will be collected with the Female Sexual Function Questionnaire Index. The highest score that can be obtained from the scale is 45, and as the total score decreases, it is considered as a decrease in sexual function.
Sexual function-fourth evaluation | 6 month after surgery
  Sexual function will be evaluated 4 times in the postoperative period.Data will be collected with the Female Sexual Function Questionnaire Index. The highest score that can be obtained from the scale is 45, and as the total score decreases, it is considered as a decrease in sexual function.
Sexual Quality of Life--first evaluation | before surgery
  Sexual quality of life will be evaluated 4 times in the perioperative period.Data will be collected with the Sexual Life Quality Scale-Female (CYKÖ-K). The score that can be obtained from the scale is between 18-108. A high score from the scale indicates that the quality of sexual life is good.
Sexual Quality of Life--second evaluation | 1 month after surgery
  Sexual quality of life will be evaluated 4 times in the perioperative period.Data will be collected with the Sexual Life Quality Scale-Female (CYKÖ-K). The score that can be obtained from the scale is between 18-108. A high score from the scale indicates that the quality of sexual life is good.
Sexual Quality of Life--third evaluation | 3 month after surgery
  Sexual quality of life will be evaluated 4 times in the perioperative period.Data will be collected with the Sexual Life Quality Scale-Female (CYKÖ-K). The score that can be obtained from the scale is between 18-108. A high score from the scale indicates that the quality of sexual life is good.
Sexual Quality of Life--fourth evaluation | 6 month after surgery
  Sexual quality of life will be evaluated 4 times in the perioperative period.Data will be collected with the Sexual Life Quality Scale-Female (CYKÖ-K). The score that can be obtained from the scale is between 18-108. A high score from the scale indicates that the quality of sexual life is good.

SECONDARY OUTCOMES:
Fear of sexual activity-first evaluation | before surgery
  Fear of sexual activity will be evaluated 4 times in the perioperative period.The patient's fear of sexual activity will be evaluated with the VAS. The scale has "no fear" at the left end (0) and "most intense fear possible" at the right end (10). A high score from the scale indicates a high level of fear, while a score of 0 indicates that there is no fear.
Fear of sexual activity-second evaluation | 1 month after surgery
  Fear of sexual activity will be evaluated 4 times in the perioperative period.The patient's fear of sexual activity will be evaluated with the VAS. The scale has "no fear" at the left end (0) and "most intense fear possible" at the right end (10). A high score from the scale indicates a high level of fear, while a score of 0 indicates that there is no fear.
Fear of sexual activity-third evaluation | 3 month after surgery
  Fear of sexual activity will be evaluated 4 times in the perioperative period.The patient's fear of sexual activity will be evaluated with the VAS. The scale has "no fear" at the left end (0) and "most intense fear possible" at the right end (10). A high score from the scale indicates a high level of fear, while a score of 0 indicates that there is no fear.
Fear of sexual activity-fourth evaluation | 6 month after surgery
  Fear of sexual activity will be evaluated 4 times in the perioperative period.The patient's fear of sexual activity will be evaluated with the VAS. The scale has "no fear" at the left end (0) and "most intense fear possible" at the right end (10). A high score from the scale indicates a high level of fear, while a score of 0 indicates that there is no fear.
satisfaction with sexual activity-first evaluation | before surgery
  satisfaction with sexual activity will be evaluated 4 times in the perioperative period.The patient's satisfaction with sexual activity will be evaluated with the VAS. At the left end of the scale, "I am not satisfied at all" is written, and at the right end (10) "Highest possible satisfaction" is written. A high score from the scale indicates a high level of satisfaction, while a score of 0 indicates dissatisfaction.
satisfaction with sexual activity-second evaluation | 1 month after surgery
  satisfaction with sexual activity will be evaluated 4 times in the perioperative period.The patient's satisfaction with sexual activity will be evaluated with the VAS. At the left end of the scale, "I am not satisfied at all" is written, and at the right end (10) "Highest possible satisfaction" is written. A high score from the scale indicates a high level of satisfaction, while a score of 0 indicates dissatisfaction.
satisfaction with sexual activity-third evaluation | 3 month after surgery
  satisfaction with sexual activity will be evaluated 4 times in the perioperative period.The patient's satisfaction with sexual activity will be evaluated with the VAS. At the left end of the scale, "I am not satisfied at all" is written, and at the right end (10) "Highest possible satisfaction" is written. A high score from the scale indicates a high level of satisfaction, while a score of 0 indicates dissatisfaction.
satisfaction with sexual activity-fourth evaluation | 6 month after surgery
  satisfaction with sexual activity will be evaluated 4 times in the perioperative period.The patient's satisfaction with sexual activity will be evaluated with the VAS. At the left end of the scale, "I am not satisfied at all" is written, and at the right end (10) "Highest possible satisfaction" is written. A high score from the scale indicates a high level of satisfaction, while a score of 0 indicates dissatisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice ÖNER CENGİZ, Study Director — Ankara University
Locations (1):
- Hatice ÖNER CENGİZ, Altındağ, Ankara, Turkey (Türkiye)